CLINICAL TRIAL: NCT00238498
Title: A Clinical Study to Assess the Efficacy and Safety of Vildagliptin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A1202
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
This study was not conducted in the United States. The purpose of this study was to assess the safety and effectiveness of a number of doses of vildagliptin, an unapproved drug, in the treatment of people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Patients who have been placed on diet and exercise therapy without achievement of glycemic control
* Outpatients

Exclusion Criteria:

* Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes
* Significant cardiovascular diseases
* Significant diabetic complications
* Other protocol-defined exclusion criteria may apply

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2004-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 12 weeks

SECONDARY OUTCOMES:
Change from baseline for postprandial glucose at 12 weeks
Change from baseline on fasting plasma glucose at 12 weeks
Change from baseline on postprandial glucose AUC at 12 weeks
Change from baseline in HOMA B at 12 weeks
Change from baseline in HOMA IR at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals